CLINICAL TRIAL: NCT03518164
Title: A Randomized, Prospective Clinical Trial Comparing the Use of Allograft Bone With Autograft Iliac Crest Bone in Anterior Cervical Spine Fusion Surgeries
Brief Title: Comparing Allograft to Autograft Bone in ACDF Surgeries
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator stopped study
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Robert F. Heary, MD, Professor, Neurosurgery, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20170000404
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Myelopathy
MeSH Terms: conditions — Spinal Cord Diseases | interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allograft (Other): Bone graft
  Interventions: Procedure: Allograft
- Autograft (Other): Bone from iliac crest
  Interventions: Procedure: Allograft

INTERVENTIONS:
Procedure: Allograft — Bone graft

SUMMARY:
Anterior cervical discectomy and fusion (ACDF) is a surgery performed from the front of the neck in which damaged discs are removed and a bone graft is inserted into the space to allow the bone to grow together to set up a bridge or fusion between the bones of the spine. The purpose of this study is to determine whether there is an advantage to using autograft (bone material taken from the patient's own hip) or allograft (bone material derived from other sources) when performing ACDF. Both of these materials are routinely used by surgeons in ACDF surgeries. Neither is experimental.

Subjects who participate in this study will be randomized to receive either allograft or autograft bone for the surgery. They will receive the 2 level ACDF surgeries routinely employed by the surgeons. The same screw-plate fixation will be used for all subjects in the trial and the same allograft material will be used for all subjects who are randomized to the allograft arm of this study.

A determination will be made as to whether there is a difference in fusion rates associated with the choice of either allograft bone or autograft bone based on the subjects' x-rays one year post surgery. The study will also determine whether there are differences in clinical and functional outcomes associated with the choice of bone graft as measured by patient-reported outcomes instruments collected. In addition, the study will examine whether there are differences in clinical and radiographic outcomes based on choice of bone graft for the subgroup of smokers participating in the study. Overall hospitalization costs will also be obtained and compared as an indication as to whether one method or the other may be superior from a financial standpoint.

DETAILED DESCRIPTION:
The study is a prospective, randomized multicenter trial. Approximately 200 subjects will be enrolled at 12 sites throughout the United States and Canada. Up to 250 subjects may be enrolled to account for screen failures. Rutgers, New Jersey Medical School is the coordinating center for the study. The purpose of this study is to determine whether there is an advantage to using autograft (bone material taken from the patient's own hip) or allograft (bone material derived from other sources) when performing ACDF. Both of these materials are routinely used by surgeons in ACDF surgeries. Neither is experimental.

Using a computer randomization program, the central study coordinating site will randomize subjects in a 1:1 ratio to either the autograft or allograft arm of the trial. Surgery is then scheduled in the routine manner. The same ACDF surgeries routinely employed by study surgeons will be performed with screw-plate fixation using the same Medtronic system for all surgeries. In addition, all surgeons will use the same allograft struts, also be provided by Medtronic [Cornerstone].

Postoperative management will be the usual and customary procedures followed by the spine surgeons participating in the trial. This would include a wound check at some point in the first two weeks following discharge with clinical and radiographic studies performed at 6 weeks, 3 months, 6 months, 1 year, and 2 years after the index surgery. Baseline and 1 year postoperative X-rays will be collected for the study. As the "gold standard" for the evaluation of fusion is the presence of bridging trabecular bone across an intended fusion interspace as well as the lack of motion between the spinous processes at the treated levels, dynamic plain film radiographs in neutral, flexion and extension will be obtained to determine fusion status. Neuroradiologists will review the subjects' 1 year radiographs. If these images are unable to definitively clarify whether a fusion has occurred at the 1 year time point, then CT scan examinations would be obtained as standard of care to make the determination. Review of these CT scans for the trial would also be performed by a blinded study radiologist. Sagittal and coronal reconstructed views will be generated. All subjects' imaging studies will be reviewed by a Board certified radiologist certified in neuroradiology. The flexion and extension cervical spine radiographs would be obtained to determine motion between the spinous processes and the presence of bridging trabecular bone. This will include preoperative and postoperative (1 year) imaging in which the neuroradiologist will be blinded to the readings of any outside radiologists or surgeons. At 1 year, the neuroradiologist will provide a binomial response of either "fused" or "not fused". Partial fusions will be considered not fused for the purposes of this study. The decision of the blinded neuroradiologist will be final regardless of the surgeon's impressions of the imaging studies.

Subject visits will occur at the patients' standard of care clinical visits at baseline/screening and at 6 weeks, 3 months, 6 months, 1 year and 2 years post-surgery. Study questionnaires and routine physician evaluations will be completed at each of these visits. X-rays will be collected and reviewed at the baseline and 1 year visits. A CT scan will be collected at 1 year only in the event that radiographs cannot determine whether fusion has occurred. Subjects will be monitored for adverse events at each visit.

Complications related to the cervical and the iliac regions will be carefully observed. In the cervical spine, the complications would include: persistent neck pain, persistent arm pain, new neurological findings, instrumentation failure, fusion failure, dysphagia, and voice issues (hoarseness and/or weakness). Specific to the iliac patients, complications related to pain, bleeding, infection, development of meralgia paresthetica, pelvis fracture, or other findings related to the iliac harvest would be catalogued. If reoperation is necessary, this will be recorded on a Report of Second Cervical Surgery as well the reason for the reoperation. Complications such as graft dislodgement, extrusion, or collapse will be noted. Instrumentation failure resulting in screw and/or plate fracture will be recorded. Reoperations for any reason will be identified and specific observation will be made as to whether a pseudoarthrosis was present as the rationale for the reoperation. In addition, clarification as to whether surgery was needed for an adjacent segment issue next to a previously successful fusion will be documented.

Due to concerns with swallowing dysfunction following anterior cervical surgery, all patients in the study will be evaluated prior to the surgery and at routine follow-up time points with the Dysphagia Short Questionnaire (DSQ).

Smokers will be included in the study and their patient-reported status with respect to the level of use of nicotine containing products will be documented at each visit. All smokers will be encouraged to quit smoking prior to the surgeries.

Both disease- specific and general patient outcomes will be analyzed at regular intervals. Outcomes related to neck pain, arm pain, and neurological abnormalities will be assessed. The following patient-reported outcomes measures will be administered to subjects prior to surgery and at 6 weeks, 3 months and 6 months, 1 year and 2 years: DSQ, PROMIS-PF, EQ-5D-5L, NDI, and VAS (arm and neck and iliac crest-if applicable).

ELIGIBILITY:
Inclusion Criteria:

1. Only two level anterior cervical discectomy surgeries will be considered. Indications for surgery can be myelopathy, radiculopathy, or mechanical neck pain resulting from instability. Patients for this study are individuals who would be undergoing surgery regardless of the clinical study.
2. Age between 18 and 80 years.

Exclusion Criteria:

1. Patients who have previously undergone cervical spine surgery, of any kind, will not be permitted to enroll in this study.
2. Patients who require only 1 level of surgery or who require surgery for 3 or more levels may not be enrolled.
3. Surgical issues excluding a patient from enrollment include the need for a corpectomy or the presence of opacification of the posterior longitudinal ligament (OPLL).
4. Patients requiring regular usage of glucocorticoid medications, for any reasons (rheumatological, pulmonary, immunological, endocrinological, etc.) will be excluded.
5. Patients taking non-steroidal anti-inflammatory (NSAID) medications would be required to discontinue their medications 10 days prior to the date of surgery and for a minimum of 6 weeks following surgery. If the patient is unable or unwilling to do this, then that patient would be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Smoking survey | 2 years
  smoking

CONTACTS AND LOCATIONS:
Overall Officials: Robert F. Heary, MD, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: No